CLINICAL TRIAL: NCT06525285
Title: Modified Coronally Advanced Flap and Enamel Matrix Derivative With and Without Connective Tissue Graft Wall Technique for the Treatment of Class III and IV Gingival recessions-a Randomized Control Trial
Brief Title: MCAF and EMD With and Without CTG Wall Technique for the Treatment of Class III and IV Gingival recessions-a Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_147464
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Connective tissue graft wall technique
  Interventions: Procedure: Connective tissue graft wall technique
- Control group (Active Comparator): Connective tissue graft
  Interventions: Procedure: Connective tissue graft wall technique

INTERVENTIONS:
Procedure: Connective tissue graft wall technique — Harvested connective tissue graft will be placed over the exposed root surface like a wall to cover the gingival recession
  Other Names: Connective tissue graft technique

SUMMARY:
Research is to compare and evaluate the clinical outcomes of the Connective tissue graft wall technique with modified coronally advanced flap to improve root coverage and clinical attachment levels in Miller's class III and IV gingival recession.

DETAILED DESCRIPTION:
Research is to compare and evaluate the clinical outcomes of the Connective tissue graft wall technique with modified coronally advanced flap to improve root coverage and clinical attachment levels in Miller's class III and IV gingival recession. The objectives is to assess the probing pocket depth reduction, clinical attachment level gain, patient esthetic evaluation, complete root coverage and mean root coverage. the control group will be treated with modified coronally advanced flap with connective tissue graft and enamel matrix derivative and the study group will be treated with modified coronally advanced flap with connective tissue graft wall and enamel matrix derivative. The total number of participants included will be 24 (Control-12; Study-12) with a 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-60 years
* Systemically healthy individuals
* Participants with Miller's Class III and IV or Cairo's RT3 gingival recession in maxillary and mandibular anteriors.
* Participants with Nordland and Tarnow's papillary recession of either I, II or III.
* Presence of interdental PPD, CAL and recession
* Radiographic evidence of interdental bone loss
* No prior experience of root coverage procedures
* Able to achieve good oral hygiene and control gingivitis in the whole of the dentition (FMPS < 25% and FMBS < 25%).

Exclusion Criteria:

* Grade III mobile teeth
* Pathologically migrated teeth
* Endodontically treated teeth
* Open contacts
* Pregnancy and lactating women
* Participants with systemic conditions
* Untreated periodontitis
* Persistence of uncorrected gingival trauma from tooth brushing
* Self-reported current smoking
* Presence of medical contraindications to elective surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-19 (Estimated); Primary Completion 2025-01-12 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Root coverage | 6 months
  Mean root coverage Cairo's RT3 gingival recession treated with MCAF + CTG wall + EMD technique is non-inferior to MCAF + CTG + EMD in terms of root coverage.

SECONDARY OUTCOMES:
Gingival health and evaluation | 6 months
  clinical attachment level

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Prabhuji MLV, Bengaluru, Karnataka, India